CLINICAL TRIAL: NCT05548309
Title: The Effect of High Flow Nasal Cannula Versus Simple Face Mask Oxygen Therapy on Pulmonary Complications After Major Abdominal Surgeries
Brief Title: HFNC Versus Oxygen Face Mask on Postoperative Pulmonery Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Huda abdellatif Boghdady, assistant lecturer,alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: High Flow Nasal cannula
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Post Operative Pulmonary Complications
Keywords: HFNC; Pulmonary complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula (Active Comparator): High flow nasal cannula (HFNC) was inserted through nasal prongs (Fisher & Paykel Healthcare, Auckland, New Zealand) . FiO2 was continuously measured by a dedicated system (AIRVO™ 2; Fisher & Paykel Healthcare, Auckland, New Zealand) .
  Interventions: Device: HFNC
- oxygen face mask (Active Comparator): Simple oxygen face mask was applied to patients starting with flow rate 6L/min .
  Interventions: Device: Oxygen face mask

INTERVENTIONS:
Device: HFNC — High flow nasal cannula (HFNC) was inserted through specific medium/large nasal prongs . FiO2 was continuously measured by a dedicated system (AIRVO™ 2; Fisher & Paykel Healthcare, Auckland, New Zealand) connected to the HFNC. Starting flow 35 L/min, temperature 31oc. The flow was titrated up to 60L/min with a target SpO2 of ≥94%.
  Arms: High flow nasal cannula
Device: Oxygen face mask — Oxygen face mask was applied to patients postoperatively with starting flow 8L/min and titration of flow up to 10 L/min with target SpO2 of ≥94%
  Arms: oxygen face mask

SUMMARY:
Eighty adult patients were randomly categorized into two equal groups (forty patients each): HFNC was applied to group I, and a simple oxygen face mask was applied to group II. Postoperative pulmonary complications were assessed for five days later.

DETAILED DESCRIPTION:
After an informed written consent taken from all the patients included in this study, they were assessed thoroughly by:

* Detailed medical and surgical history taking.
* Complete clinical examination.
* Routine laboratory investigations, including complete blood picture, blood urea nitrogen, serum creatinine, prothrombin (PT), activated partial thromboplastin (aPTT) times, thrombin time, fasting blood sugar.
* Electrocardiograph (ECG) and chest x-ray.

On arrival of the patient to the operative theatre peripheral intravenous cannula gauge 18 was inserted and all patients were attached to multichannel monitor (CARESCAPE™ Monitor B650) to display the following:

1. Heart rate (beats/ minute).
2. Non-invasive systolic, diastolic, and mean arterial blood pressure (mmHg).
3. Respiratory rate (breaths/min).
4. Peripheral oxygen saturation (%).
5. End tidal carbon dioxide (mmHg). Epidural catheter was inserted for all patients at level T7-T9, loading dose 1-1.5 ml/segment of 0.125% bupivacaine with fentanyl 1mic/ml and was continued as an infusion intraoperatively combined with general anaesthesia with infusion rate 5ml/hour. Mechanical ventilation was initiated after tracheal intubation using volume control mode.

At the end of the surgery lung recruitment was done by closing an adjustable pressure-limiting valve at continuous positive airway pressure 30 cmH2O2 for 30 seconds.Extubation was done after patients fulfilling the criteria of extubation.

Oxygen therapy was delivered through simple face mask while transportation to ICU with flow rate 6-10L/min titrated to maintain SpO2 ≥ 94%.

Patients were randomly categorized using closed envelope technique into 2 equal groups (40 patients each as calculated by the department of biomedical informatics and medical statistics, medical research institute, Alexandria University) Group I: High flow nasal cannula (HFNC) was inserted through specific medium/large nasal prongs (Fisher & Paykel Healthcare, Auckland, New Zealand). FiO2 was continuously measured by a dedicated system (AIRVO™ 2; Fisher & Paykel Healthcare, Auckland, New Zealand) connected to the HFNC. Starting flow 35 L/min, temperature 31oc. the flow was titrated up to 60L/min with a target SpO2 of ≥94%.

Group II: Simple oxygen face mask was applied to patients starting flow rate 6L/min and titration of flow rate up to 10L/min was done to target peripheral oxygen saturation SpO2 of ≥94%.

Gradual weaning started after 6 hours when satisfactory ABG obtained, targeting SpO2 ≥ 94%.Oxygen therapy was discontinued and noninvasive positive pressure ventilation (NIPPV) was started for both groups when patients developed moderate acute hypoxemic respiratory failure at least 2 of the following criteria were met:

1. Respiratory frequency more than 25 and less than 35 breaths/min persistent for at least 1 hour.
2. Clinical signs of respiratory distress (dyspnea, significant use of accessory muscles, or paradoxical abdominal motion).
3. Respiratory acidosis (PH less than 7.35 units and PaCO2 more than 45 mm Hg).
4. Moderate hypoxemia defined as PaO2/FiO2 more than 150 and less than 300.

Endotracheal intubation was performed when the patients of both groups developed severe acute hypoxemic respiratory failure (at least 2 of the following criteria) were met:

1. Respiratory frequency 40 breaths/min.
2. Clinical signs of respiratory distress (dyspnea, significant use of accessory muscles, or paradoxical abdominal motion).
3. Respiratory acidosis with an arterial PH less than 7.30, and PaCO2 more than 45 mm Hg).
4. Severe hypoxemia defined as PaO2/FiO2 less than 150. All other treatments were continued according to the standard care in ICU with patients of both groups receiving physiotherapy, upright positioning, incentive spirometry, and early mobilization.

Incidence of postoperative pulmonary complications detected in ICU by daily chest x-ray and lung US .

Chest X-ray was done on day 1, day3, day 5 and the incidence of postoperative pulmonary complications were recorded according to European Perioperative Clinical Outcome definitions (EPCO).

Lung ultrasound using (Sonosite M-Turbo® Ultrasound System) linear transducer (L38Xi 10-5 MHZ) was performed on postoperative day (POD) 0, day1, day2, day3, day4, day5, lung ultrasound views were obtained according to the Bed Side Lung Ultrasound in Emergency protocol (BLUE).

Two hands placed this way (size equivalent to the patient's hands, upper hand touching the clavicle, thumbs excluded) correspond to the location of the lung, and allow three standardized points to be defined .

1. The upper BLUE point is in the middle of the upper hand. 2. The lower BLUE point is in the middle of the lower palm. 3. The poster lateral alveolar or pleural syndromes (PLAPS) point is defined by the intersection of a horizontal line at the level of the lower BLUE point and a vertical line at the posterior axillary line.BLUE profile for each BLUE point and BLUE profile per hemi thorax will be determined as follows:

1. The A profile associates anterior lung sliding with A lines .
2. The A' profile is an A profile with abolished lung sliding.
3. The B profile predominantly multiple (>2) anterior diffuse B lines indicating interstitial syndrome associates anterior lung sliding .
4. The B' profile is a B-profile with abolished lung sliding.
5. The C profile indicates anterior lung consolidation, regardless of size and number, thickened, irregular pleural line is an equivalent.
6. The A/B profile is a half A profile at one lung, a half B profile at another. Furthermore, the postero lateral alveolar and/or pleural syndrome (PLAPS) was determined at PLAPS point and was scored as positive or negative. When consolidation and/or pleural effusion were detected they were scored separately; for differentiation between pneumonia and atelectasis, fever, leukocyte count, and C-reactive protein were looked for.Diaphragmatic excursion was measured (On admission day 0, day1, day 2, day3, day4, day5).

The low frequency curvilinear transducer (C60xi 5-2 MHZ) was placed in bilateral costal margins between the anterior and posterior axillary lines for longitudinal scanning. Images of diaphragmatic excursions was obtained using the liver and spleen as acoustic windows during full respiration. With normal breathing of patients in the 45° semi supination position, the maximum vertical axis between the adjacent peaks and valleys using the sinusoid in the M mode was measured as the diaphragmatic excursion movement .

Multiple respiratory cycles of at least three cycles were recorded and the average was taken. Every side measurements (right and left hemidiaphragms) was measured and calculated separately and then the average of measurements of the two sides were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (50-70 years).
* Patients with American Society of Anesthesiologists (ASA) status I-III.
* Patients with body mass index less than 35kg/m2.
* Patients scheduled for major elective upper abdominal surgeries (gastrectomy, hepatic resection, pancreatectomy, Whipple procedures,..).
* Upper abdominal surgery with an abdominal incision longer than 5 cm that is above or extending above the umbilicus.
* Upper abdominal surgeries with an anticipated duration of two hours or more.

Exclusion Criteria :• Patients who refuse to participate in the study.

* Patients with tracheostomy

  .• Patients with pre-existing pulmonary disease (pleural effusion, pneumothorax or pulmonary atelectasis).
* Patients with pre-existing obstructive sleep apnea.
* Patients with any nasal or facial defect that could impede use of HFNC (Nasal septal defect or any form of facial deformity).
* Impaired consciousness Glasgow coma scale (GCS) less than 12.
* Hemodynamic instability as systolic blood pressure less than 90 mmHg, mean arterial blood pressure less than 65 mmHg or vasopressor requirement.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
To compare the effect of HFNC and simple face mask oxygen therapy regarding postoperative pulmonary complications within five days after major elective upper abdominal surgeries. | 5 days postoperatively
  postoperative pulmonery complications detected by lung ultrasound and chest x-ray

SECONDARY OUTCOMES:
To detect the need for escalation of respiratory support | 5 days postoperatively
  The need to non invasive ventilation or intubation
Intensive care unit length of stay(days) | 14 days postoperatively
  Discharge criteria from ICU to ward included: Toleration of mobilization, absence of vasoactive treatment, stable hemodynamic, satisfactory respiratory conditions, unnecessary for invasive monitoring, and no further active interventions planned
Hospital length of stay(days) | 21 days postoperatively
  The criteria for hospital discharge included: the presence of sinus rhythm, absence of pyrexia and wound infection, normal routine blood tests, satisfactory chest X-ray, and full mobility

CONTACTS AND LOCATIONS:
Overall Officials: Dorya fekry, MD, Study Director — Alexandria University; Ahmed EL-Attar, MD, Study Director — Alexandria University; Mohamed El Hadidy, MD, Study Director — Alexandria University
Locations (1):
- Alexandria University,Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
clinical trial
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one month